CLINICAL TRIAL: NCT05146583
Title: Injection of Autologous Bone Marrow Aspirate in Patients With Degenerative Disc Disease: a Phase I Clinical Trial
Brief Title: Injection of Autologous Bone Marrow Aspirate in Patients With Degenerative Disc Disease.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: New York Presbyterian Hospital (Other)
Responsible Party: Principal Investigator, Pravesh Gadjradj, on behalf of PI: Prof.dr.R.Hartl, chief of spine surgery, New York Presbyterian Hospital
Other Study IDs: NYP19-04020103
Record Dates: First submitted 2021-11-10; First posted 2021-12-07 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Lumbar Disc Disease
Keywords: Sciatica; Lumbar Disc Herniation; Discectomy
MeSH Terms: conditions — Intervertebral disc disease; Sciatica; Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Autologous bone marrow aspirate injected intradiscal after microdiscectomy — Harvested from SI-joint, 2-5ml BMA is injected in the discectomy defect.
Procedure: Discectomy only — Transflaval discectomy with or without the use of a microtube (according to surgeons' preference).

SUMMARY:
Lumbar discectomy and injection of purified cellular bone marrow concentrate or lumbar discectomy only

DETAILED DESCRIPTION:
In order to find a regenerative treatment for back pain from DDD, cell based therapies have become of increasing interest. Recent clinical studies have shown promising improvement in pain and disc hydration, thus indicating a regenerative effect.

The use of mesenchymal stem cells for regeneration of degenerated connective tissue of mesenchymal origin has proven efficient in multiple recent studies. However, the acquisition of mesenchymal stem cells (MSC) is always an extensive procedure requiring either enzymatic or genetic manipulation of acquired tissues. Thus, the use of these MSCs is highly controversial and raises concerns in terms of patient safety.

One of the most commonly used sources for MSCs is bone marrow tissue. Even when not manipulated, these tissues already contain a significant amount of mesenchymal stem cells and growth factors. Therefore, they are used for regenerative treatments of multiple degenerative musculoskeletal diseases.

This is an exploratory pilot study which aims to compare patient outcomes between two treatments approaches for DDD that are currently being used in clinic. While micro- discectomy is the standard of care for DDD, micro-discectomies with autologous bone marrow cell injections have been used in clinic in the past year. The goal of this study is to determine if the bone marrow injection group is superior compared to the control group (state of the art micro-discectomies) in enhancing degenerative disc recovery and improving or preventing back pain.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥18 years of age
2. Radiologically (MRI) confirmed diagnosis degenerative disc disease of the lumbar spine and/or lumbar disc herniation
3. Unresponsive to conservative/non-operative treatment for >3 months
4. Psychosocial, mental and physical ability to understand and to adhere to this protocol, especially adhering to the visit schedule follow-ups, and observe treatment plan
5. Signed and dated informed consent document prior to any study-related procedures indicating that the patient has been informed of all pertinent aspects of the trial study-related procedures

Exclusion Criteria:

1. Pregnant or breastfeeding patients
2. Active malignancy
3. Active chronic or acute infection
4. Autoimmune disorder that impacts the lumbar spine (Ankylosing spondylitis, lupus eg.)
5. Acute Episode or major mental illness
6. Major cognitive impairment causing to inability to understand informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic lumbar disc herniation and discogenic back pain who meet the inclusion criteria may be eligible for this procedure.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Numeric Rating for Back pain at 12 months | Baseline, 3 months, 6 months, 12 months after surgery
  0 to 10 NRS

SECONDARY OUTCOMES:
Change in Oswestry Disability Index at 12 months | Baseline, 3 months, 6 months, 12 months after surgery
  0 to 100 PROM to measure low back disfunction
Disc Height Index | Baseline and 12 months or longer folllow-up after surgery
  MRI measurement
Pfirrman grading | Baseline and 12 months or longer folllow-up after surgery
  MRI measurement
Change in NRS Leg pain | Baseline, 3 months, 6 months, 12 months after surgery
  0 to 10 NRS
Complications | Continrous monitoring during study during one year after surgery
  Infections, reoperations, blood loss.

CONTACTS AND LOCATIONS:
Locations (1):
- New York Presbytarian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No